CLINICAL TRIAL: NCT00785291
Title: A Randomized Phase III Trial of Weekly Paclitaxel Compared to Weekly Nanoparticle Albumin Bound Nab-paclitaxel or Ixabepilone With or Without Bevacizumab as First-Line Therapy for Locally Recurrent or Metastatic Breast Cancer
Brief Title: Paclitaxel, Nab-paclitaxel, or Ixabepilone With or Without Bevacizumab in Treating Patients With Stage IIIC or Stage IV Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00476; NCI-2009-00476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CTSU 40502; CDR0000617539; NCCTG N063H; CALGB-40502; PCALGB-40502_A11PAMDREVW01; CALGB 40502 (Other: Alliance for Clinical Trials in Oncology); CALGB-40502 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; HER2/Neu Positive; Progesterone Receptor Negative; Progesterone Receptor Positive; Recurrent Breast Carcinoma; Stage IIIC Breast Cancer AJCC v6; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; ixabepilone; Epothilones; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Paclitaxel) (Active Comparator): Patients receive 90 mg/m^2 paclitaxel IV over 1 hour on days 1, 8, and 15. Patients may receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Questionnaire Administration
- Arm B (Nab-paclitaxel) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Patients may also receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Nab-paclitaxel; Other: Questionnaire Administration
- Arm C (Ixabepilone) (Experimental): Patients receive ixabepilone IV over 60 minutes on days 1, 8, and 15. Patients may also receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15. (closed to accrual as of 7/18/11)
  Interventions: Biological: Bevacizumab; Drug: Ixabepilone; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Zirabev
Drug: Ixabepilone — Given IV
  Other Names: (1S,3S,7S,10R,11S,12S,16R)-7,11-Dihydroxy-8,8,10,12,16-pentamethyl-3-[(1E)-1-methyl-2-(2-methyl-4-thiazolyl)ethenyl]-17-oxa-4-azabicyclo[14.1.0]heptadecane-5,9-dione; Azaepothilone B; BMS 247550; BMS-247550; BMS247550; Epothilone; Epothilone-B BMS 247550; Ixempra
  Arms: Arm C (Ixabepilone)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
  Arms: Arm B (Nab-paclitaxel)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm A (Paclitaxel)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies the side effects and how well different chemotherapy regimens with or without bevacizumab work in treating patients with stage IIIC or stage IV breast cancer. Drugs used in chemotherapy, such as paclitaxel, paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel), and ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab may block tumor growth by targeting certain cells and slowing the growth of blood vessels to the tumor. It is not yet known which treatment regimen is more effective in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival (PFS) in patients with metastatic breast cancer receiving nab-paclitaxel versus paclitaxel (control arm).

II. To compare PFS in patients receiving ixabepilone versus paclitaxel.

SECONDARY OBJECTIVES:

I. To compare the objective response rate, duration of response, and time to treatment failure in patients receiving nab-paclitaxel versus paclitaxel, and to separately compare these endpoints in patients receiving ixabepilone versus paclitaxel.

II. To compare the 12-month rate of progression in patients receiving nab-paclitaxel versus paclitaxel, and to separately compare this endpoint in patients receiving ixabepilone versus paclitaxel.

III. To determine toxicities in patients receiving nab-paclitaxel as compared to paclitaxel, and in patients receiving ixabepilone as compared to paclitaxel.

IV. To compare overall survival in patients receiving nab-paclitaxel versus paclitaxel, and to separately compare overall survival in patients receiving ixabepilone versus paclitaxel.

V. To evaluate the relationships between secreted protein, acidic, cysteine-rich (SPARC) overexpression and changes in blood levels of caveolin-1 (Cav-1) to PFS and secondary endpoints of response during treatment with nab-paclitaxel as compared to paclitaxel, and with ixabepilone as compared to paclitaxel.

VI. To evaluate the relationships between changes in blood levels of circulating tumor cells (CTCs) and circulating endothelial cells (CECs) to PFS and secondary endpoints of response during treatment with nab-paclitaxel as compared to paclitaxel, and with ixabepilone as compared to paclitaxel.

VII. To evaluate the association of expression levels of the microtubule associated proteins tau and beta-tubulin isotype composition with PFS and secondary endpoints of response during treatment with nab-paclitaxel as compared to paclitaxel, and with ixabepilone as compared to paclitaxel.

VIII. To investigate a potential cytochrome P450, family 2, subfamily C polypeptide 8, 2, 3 (CYP2C8*2/*3) by paclitaxel interaction with respect to progression-free survival (PFS).

IX. To determine if CYP2C8*2 and CPY2C8*3 are associated with paclitaxel-induced peripheral neuropathy.

X. To perform exploratory analysis of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4), cytochrome P450, family 3, subfamily A, polypeptide 5 (CYP3A5), ATP-binding cassette, sub-family B (MDR/TAP), member 1 (ABCB1) and ATP-binding cassette, sub-family C (CFTR/MRP), member 2 (ABCC2) polymorphisms with response and toxicity profiles.

XI. To prospectively collect data on sociodemographics, non-cancer morbidities, and receipt of post-trial therapy to evaluate the role of potential disparities on survival from cancer.

XII. To evaluate the relationship between physical activity behaviors at the time of enrollment in the protocol and progression-free and overall survival.

XIII. To identify baseline factors that predict the risk of grade 3, 4, or 5 toxicity in patients receiving treatment with weekly paclitaxel, nab-paclitaxel, or ixabepilone combined with or without bevacizumab.

XIV. To perform an exploratory analysis of whether other factors included in patient assessments (either individually or in combination) predict the risk of grade 3, 4, or 5 toxicity in patients receiving weekly paclitaxel, nab-paclitaxel, or ixabepilone combined with or without bevacizumab, with a specific focus on the relationship between pre-existing hypertension or neuropathy.

XV. To compare the associations of baseline factors to grade 3, 4, or 5 toxicity in patients receiving weekly paclitaxel, nab-paclitaxel, or ixabepilone combined with or without bevacizumab.

XVI. To explore whether longitudinal changes in factors are in association with the occurrence of grade 3, 4, or 5 toxicities in patients with weekly paclitaxel, nab-paclitaxel, or ixabepilone combined with or without bevacizumab.

XVII. To explore the association between grade 2-4 neuropathy and longitudinal changes in the following functional status measures: a) Older Americans Resources and Services (OARS) Multidimensional Functional Assessment Questionnaire (MFAQ) (Instrumental Activities of Daily Living [IADL]); b) Medical Outcomes Study (MOS) Physical Functioning; c) Karnofsky Performance Status Rated Healthcare Professional; d) Timed "Up and Go"; e) OARS Physical Health Section.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A (WEEKLY PACLITAXEL): Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15. Patients may also receive bevacizumab IV over 30-90 minutes on days 1 and 15.

ARM B (WEEKLY NAB-PACLITAXEL): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Patients may also receive bevacizumab as in Arm A.

ARM C (WEEKLY IXABEPILONE): Patients receive ixabepilone IV over 60 minutes on days 1, 8, and 15. Patients may also receive bevacizumab as in Arm A. (closed to accrual as of 7/18/11)

In all arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 6 months for 2 years and then annually for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of invasive cancer of the breast
* Stage IV disease or stage IIIC disease (using American Joint Committee on Cancer [AJCC] criteria, 6th edition) not amenable to local therapy
* Patients may not have a "currently active" second malignancy other than non-melanoma skin cancers; patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse
* Patients with human epidermal growth factor receptor 2 (HER2) negative disease are eligible; patients with HER2+ disease are eligible providing they have previously received trastuzumab or lapatinib; documentation of progression on HER2 directed therapy is not required; Her2/neu status must be known at the time of protocol registration
* Estrogen receptor (ER) and progesterone receptor (PgR) status must be known at the time of registration; ER and/or PgR >= 1% cells will be considered positive
* Prior treatment may include adjuvant or neoadjuvant taxane, however, the interval between completion of adjuvant or neoadjuvant therapy and disease recurrence must be >= 12 months
* No prior chemotherapy for metastatic breast cancer
* Any number of prior hormonal therapies are allowed; the last dose should have been administered at least 7 days prior to the initiation of protocol therapy
* Prior radiotherapy must be completed at least 2 weeks prior to study entry
* Treatment with bisphosphonates is allowed and recommended as per American Society of Clinical Oncology (ASCO) guidelines
* Prior trastuzumab or lapatinib required for patients with HER2 overexpressing tumors
* Prior treatment with bevacizumab is allowed
* Patients must not have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study registration, and must have fully recovered from any such procedure

  * The following are not considered to be major procedures: thoracentesis, paracentesis, port placement, laparoscopy, thoracoscopy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies and routine dental procedures
* Patients must not have anticipation of need for a major surgical procedure during the course of the study
* There are no restrictions on core biopsies, placement of a vascular access device or other minor procedures prior to registration

  * Placement of a vascular access device after starting study therapy should be performed between day 15 and 28 of a treatment cycle (but not less than 48 hours before the next dose of bevacizumab) to allow for sufficient healing
* Patients must have measurable disease (target lesions): measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2.0 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan

  * Lesions that are considered non-measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonitis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Patients with pre-existing peripheral neuropathy >= grade 2 are not eligible for this study
* Patients must have an Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status of =< 1 to be eligible for this trial
* Women must not be pregnant or breast feeding; premenopausal women must have a negative serum or urine beta-human chorionic gonadotropin (Hcg)
* Patients with a history of Common Terminology Criteria for Adverse Events (CTCAE) grade >= 3 hypersensitivity to paclitaxel or Cremophor® EL are not eligible
* Patients with a history of abdominal fistula, or intra-abdominal abscess within 6 months prior to study registration are not eligible
* Patients with a history of gastrointestinal (GI) perforation within 12 months prior to registration are not eligible
* Patients with a history of significant bleeding episodes (e.g., hemoptysis, upper or lower GI bleeding) within 6 months prior to registration are not eligible
* Patients must not have a history of clinically significant cardiovascular disease that includes the following:

  * Uncontrolled hypertension defined as systolic blood pressure > 150 and/or diastolic blood pressure > 90 mmHg on antihypertensive medications or any prior history of hypertensive crisis or hypertensive encephalopathy
  * History of myocardial infarction or unstable angina within past 6 months
  * New York Heart Association (NYHA) congestive heart failure grade 2 or greater
  * Symptomatic peripheral vascular disease
  * Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or arterial thrombotic events
* Patients on full dose anticoagulants must be on a stable dose of warfarin, or be on a stable dose of low molecular weight (LMW) heparin; patients receiving anti-platelet or on daily prophylactic dose aspirin are eligible, as are patients receiving stable doses of anticoagulation for atrial fibrillation
* Patients may not have a history of stroke or transient ischemic attack within 6 months prior to study registration
* Patients with a history of seizures must be well controlled with standard medication
* Patients must not have progressing or untreated central nervous system (CNS) metastases or leptomeningeal disease; patients with a history of resected brain metastases with stable magnetic resonance imaging (MRI) scans for 3 months including within 4 weeks of study start are eligible; patients with a history of gamma knife radiosurgery or whole brain radiation with stable MRI scans for 3 months including within 4 weeks of study start are eligible
* No serious, non-healing wound, ulcer or bone fracture
* Life expectancy of >= 12 weeks
* Granulocytes >= 1,500/ul
* Platelet count >= 100,000/ul
* Creatinine =< 2.0 mg/dL
* Bilirubin < 1.5 mg/dL (unless due to Gilbert's syndrome)
* Transaminases (aspartate aminotransferase [AST], alanine aminotransferase [ALT]) =< 2.5 x upper limit of normal (ULN)
* Serum or urine beta-Hcg negative in premenopausal women of child-bearing potential
* Urine protein =< 1+ protein* or urine protein: creatinine ratio (UPC) < 1

  * Patients discovered to have >= 2+ proteinuria at baseline must undergo a 24-hour urine collection that must demonstrate < 1 g of protein/24 hr or UPC ratio =< 1 to allow participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2008-10-13 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S Rugo, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (704):
- United States (703):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Yale University, New Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center - West, Boca Raton, Florida
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Florida Cancer Specialists-Gainesville Cancer Center, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Dublin Hematology Oncology Care PC, Dublin, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - MercyOne Waterloo Medical Center, Waterloo, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Advent Health - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Center for Cancer Medicine-Scarborough, Scarborough, Maine
  - Maine General Medical Center-Thayer, Waterville, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - AtlantiCare Regional Medical Center -Main Campus, Pomona, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Coney Island Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Rex Cancer Center, Raleigh, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Nash General Hospital, Rocky Mount, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center at Vidant Beaufort Hospital, Washington, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma-Lakeside, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Health System, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Coastal Cancer Center-Myrtle Beach, Myrtle Beach, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Providence Holy Family Hospital, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Stover DG, Salgado R, Savenkov O, Ballman K, Mayer EL, Magbanua MJM, Loi S, Vater M, Glover K, Watson M, Wen Y, Symmans WF, Perou C, Carey LA, Partridge AH, Rugo HS. Association between tumor-infiltrating lymphocytes and survival in patients with metastatic breast cancer receiving first-line chemotherapy: analysis of CALGB 40502. NPJ Breast Cancer. 2024 Aug 21;10(1):75. doi: 10.1038/s41523-024-00683-x. PMID 39169033
- [Derived] Quintanilha JCF, Wang J, Sibley AB, Jiang C, Etheridge AS, Shen F, Jiang G, Mulkey F, Patel JN, Hertz DL, Dees EC, McLeod HL, Bertagnolli M, Rugo H, Kindler HL, Kelly WK, Ratain MJ, Kroetz DL, Owzar K, Schneider BP, Lin D, Innocenti F. Bevacizumab-induced hypertension and proteinuria: a genome-wide study of more than 1000 patients. Br J Cancer. 2022 Feb;126(2):265-274. doi: 10.1038/s41416-021-01557-w. Epub 2021 Oct 6. PMID 34616010
- [Derived] Mehrotra S, Sharma MR, Gray E, Wu K, Barry WT, Hudis C, Winer EP, Lyss AP, Toppmeyer DL, Moreno-Aspitia A, Lad TE, Valasco M, Overmoyer B, Rugo H, Ratain MJ, Gobburu JV. Kinetic-Pharmacodynamic Model of Chemotherapy-Induced Peripheral Neuropathy in Patients with Metastatic Breast Cancer Treated with Paclitaxel, Nab-Paclitaxel, or Ixabepilone: CALGB 40502 (Alliance). AAPS J. 2017 Sep;19(5):1411-1423. doi: 10.1208/s12248-017-0101-9. Epub 2017 Jun 15. PMID 28620884
- [Derived] Rugo HS, Barry WT, Moreno-Aspitia A, Lyss AP, Cirrincione C, Leung E, Mayer EL, Naughton M, Toppmeyer D, Carey LA, Perez EA, Hudis C, Winer EP. Randomized Phase III Trial of Paclitaxel Once Per Week Compared With Nanoparticle Albumin-Bound Nab-Paclitaxel Once Per Week or Ixabepilone With Bevacizumab As First-Line Chemotherapy for Locally Recurrent or Metastatic Breast Cancer: CALGB 40502/NCCTG N063H (Alliance). J Clin Oncol. 2015 Jul 20;33(21):2361-9. doi: 10.1200/JCO.2014.59.5298. Epub 2015 Jun 8. PMID 26056183
- See also: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive." — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2008 - November 2011, a total of 799 participants were recruited.
Groups:
- Arm A (Paclitaxel): Patients receive 90 mg/m^2 paclitaxel IV over 1 hour on days 1, 8, and 15. Patients may receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment continues until progression.
- Arm B (Nab-paclitaxel): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Patients may also receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment continues until progression.
- Arm C (Ixabepilone): Patients receive ixabepilone IV over 60 minutes on days 1, 8, and 15. Patients may also receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment continues until progression. (closed to accrual as of 7/18/11)
Period: Overall Study
Arm/Group | Arm A (Paclitaxel) | Arm B (Nab-paclitaxel) | Arm C (Ixabepilone)
Started | 283 | 271 | 245
Completed | 147 | 122 | 139
Not Completed | 136 | 149 | 106
Not completed — Never began treatment | 8 | 4 | 4
Not completed — Adverse Event | 39 | 70 | 56
Not completed — Death | 7 | 4 | 3
Not completed — Withdrawal by Subject | 35 | 36 | 17
Not completed — Alternative Therapy | 12 | 6 | 7
Not completed — Complicating illness | 6 | 4 | 4
Not completed — Other Medical Reasons | 29 | 25 | 15

BASELINE CHARACTERISTICS:
Population: All randomized participants are included in baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Paclitaxel) | Arm B (Nab-paclitaxel) | Arm C (Ixabepilone) | Total
Number analyzed (Participants) | 283 | 271 | 245 | 799
Age, Customized [Number; unit: participants]
  20-29 | 2 | 2 | 1 | 5
  30-39 | 15 | 18 | 17 | 50
  40-49 | 52 | 56 | 55 | 163
  50-59 | 109 | 89 | 86 | 284
  60-69 | 74 | 74 | 68 | 216
  70-79 | 24 | 28 | 15 | 67
  80+ | 7 | 4 | 3 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 268 | 243 | 788
  Male | 6 | 3 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 15 | 13 | 47
  Not Hispanic or Latino | 252 | 239 | 221 | 712
  Unknown or Not Reported | 12 | 17 | 11 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 5
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 1 | 4
  Black or African American | 42 | 45 | 26 | 113
  White | 220 | 214 | 206 | 640
  More than one race | 1 | 1 | 2 | 4
  Unknown or Not Reported | 15 | 10 | 8 | 33
Region of Enrollment [Number; unit: participants]
  United States | 283 | 271 | 245 | 799
Prior Adjuvant Taxane [Number; unit: participants]
  Yes | 125 | 120 | 107 | 352
  No | 158 | 151 | 138 | 447
Hormone Receptor Status [Number; unit: participants]
  ER/PgR Positive | 201 | 195 | 178 | 574
  ER/PgR Negative | 82 | 76 | 67 | 225
Physician's Decision to use Bevacizumab [Number; unit: participants]
  Bevacizumab planned | 51 | 44 | 15 | 110
  Bevacizumab not planned | 8 | 4 | 8 | 20
  Bevacizumab required | 224 | 223 | 222 | 669

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the interval from registration until first disease progression, regardless of site, or death resulting from any cause, which ever occurred first. Distribution was estimated using the Kaplan Meier product-limit method. Progression is defined as a 20% increase in the sum of longest diameter of target lesions (per Response Evaluation Criteria in Solid Tumors [RECIST] criteria).
Time Frame: Time from randomization to progression or death due to any cause, whichever occurs first (up to 5 years)
Population: Participants who never began protocol treatment were excluded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Paclitaxel) | Arm B (Nab-paclitaxel) | Arm C (Ixabepilone)
Number analyzed (Participants) | 275 | 267 | 241
months | 10.97 [9.79 to 12.42] | 9.3 [8.15 to 10.45] | 7.36 [6.21 to 8.18]
Statistical Analysis 1: Comparison: Arm A (Paclitaxel) vs Arm B (Nab-paclitaxel); Stratified log-rank tests are used for the two primary comparisons of PFS within an experimental arm relative to PFS within the control arm. The family-wise error rate will be controlled at a one-sided 0.025 level. This is achieved in a 3-arm trial with a common control group by conducting the marginal log-rank tests with a one-sided α = 0.0135. Sample size calculations are based on having high power to detect a hazard ratio of 1.36, in the control arm as compared to the experimental arms; Test type: Superiority or Other; p = 0.054, Log Rank — Tests were stratified by prior taxane therapy (yes/no) and hormone receptor status (positive/negative). P-values are for a test of inferiority 2-sided and are unadjusted for multiple comparisons; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [1.00 to 1.45]
Statistical Analysis 2: Comparison: Arm A (Paclitaxel) vs Arm C (Ixabepilone); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [1.28 to 1.87]

2. Secondary Outcome: Objective Tumor Response Rate
Description: Response was defined by the Response Evaluation Criteria in Solid Tumors (RECIST). A responding participant had either a Complete Response (disappearance of all target lesions) or Partial Response (30% decrease in sum of longest diameter of target lesions).
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Paclitaxel) | Arm B (Nab-paclitaxel) | Arm C (Ixabepilone)
Number analyzed (Participants) | 275 | 267 | 241
percentage of participants | 38.2 | 34.1 | 25.6

3. Secondary Outcome: Time to Treatment Failure
Description: Time from registration until treatment failure, defined as early termination of protocol therapy for any reason, first disease progression or death without progression. Surviving participants who were failure free were censored as date last known alive and failure free. Distribution was estimated using the Kaplan Meier product-limit method.
Time Frame: Time from randomization until progression, death, or yearly termination of protocol therapy (up to 5 years)
Population: Participants who never began protocol treatment were excluded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Paclitaxel) | Arm B (Nab-paclitaxel) | Arm C (Ixabepilone)
Number analyzed (Participants) | 275 | 267 | 241
months | 6.6 [5.62 to 7.2] | 5.19 [4.83 to 5.55] | 4.93 [4.21 to 5.29]

4. Secondary Outcome: 12 Month Progression Free Survival
Description: Percentage of participants who were alive and progression free at 12 months. The 12 month progression free survival, with 95% confidence interval, was estimated using the Kaplan Meier method.
Time Frame: 12 months
Population: Participants who never began protocol treatment were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Paclitaxel) | Arm B (Nab-paclitaxel) | Arm C (Ixabepilone)
Number analyzed (Participants) | 275 | 267 | 241
percentage of participants | 45 [39 to 51] | 36 [30 to 42] | 28 [23 to 35]

5. Secondary Outcome: Overall Survival
Description: Overall survival was measured as the interval from study entry until death, from any cause, or last contact. Distribution was estimated using the Kaplan Meier product-limit method.
Time Frame: Time from randomization to death or last follow-up (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Paclitaxel) | Arm B (Nab-paclitaxel) | Arm C (Ixabepilone)
Number analyzed (Participants) | 275 | 267 | 241
months | 26.55 [23.8 to 32.9] | 23.52 [20.4 to 28.2] | 23.53 [19.9 to 25.6]
Statistical Analysis 1: Comparison: Arm A (Paclitaxel) vs Arm B (Nab-paclitaxel); Test type: Superiority or Other; p = 0.20, Log Rank — Tests were stratified by prior taxane therapy (yes/no) and hormone receptor status (positive/negative); Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.92 to 1.47]
Statistical Analysis 2: Comparison: Arm A (Paclitaxel) vs Arm C (Ixabepilone); Test type: Superiority or Other; p = 0.038, Log Rank — Tests were stratified by prior taxane therapy (yes/no) and hormone receptor status (positive/negative); Hazard Ratio (HR) = 1.28, 95% CI 2-sided [1.01 to 1.61]

ADVERSE EVENTS:
Description: Adverse event data was submitted on 774 participants (Arm A: 272, Arm B: 264, Arm C: 238)
Arm/Group | Arm A (Paclitaxel) | Arm B (Nab-paclitaxel) | Arm C (Ixabepilone)
Serious Adverse Events (participants affected / at risk) | 65/272 | 80/264 | 59/238
Other Adverse Events (participants affected / at risk) | 263/272 | 248/264 | 230/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Paclitaxel) (N=272) | Arm B (Nab-paclitaxel) (N=264) | Arm C (Ixabepilone) (N=238)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 14 (17) | 18 (22) | 12 (14)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 3 (3) | 4 (5)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Stokes-Adams syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cecum perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 6 (7) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 11 (12) | 11 (12)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 19 (21) | 21 (24)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 12 (14) | 15 (16)
Chest pain (General disorders) | 1 (1) | 2 (2) | 3 (3)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Death NOS (General disorders) | 2 (2) | 2 (2) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 2 (2) | 3 (4)
Fatigue (General disorders) | 43 (56) | 56 (64) | 40 (44)
Fever (General disorders) | 2 (2) | 7 (7) | 2 (3)
General symptom (General disorders) | 0 (0) | 2 (2) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3) | 2 (2) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Anorectal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 5 (5) | 4 (4) | 3 (3)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 3 (3) | 4 (5)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 5 (6) | 7 (7)
Salivary gland infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 5 (5) | 4 (4) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 6 (6) | 5 (5)
Uterine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 3 (4) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3)
Injury to carotid artery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intraoperative gastrointestinal injury - Teeth (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0)
ADH abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 3 (4) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 6 (7)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 2 (3) | 3 (3)
INR increased (Investigations) | 0 (0) | 2 (3) | 2 (2)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 7 (8) | 17 (19) | 7 (9)
Lymphocyte count decreased (Investigations) | 3 (3) | 2 (2) | 6 (6)
Neutrophil count decreased (Investigations) | 16 (19) | 36 (39) | 14 (16)
Platelet count decreased (Investigations) | 3 (3) | 13 (13) | 10 (10)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 5 (7) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 6 (7) | 10 (12) | 7 (7)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (7) | 8 (9) | 8 (10)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 9 (10) | 11 (12)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 9 (10) | 6 (7)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (6) | 8 (9) | 4 (4)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (5) | 5 (6) | 9 (9)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3) | 8 (9) | 7 (7)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (10) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 5 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 4 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 12 (13) | 10 (10)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 3 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (6) | 5 (6) | 5 (5)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 5 (5) | 10 (11) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 35 (45) | 43 (50) | 32 (38)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 4 (4) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (2)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 8 (9) | 10 (10) | 7 (7)
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1)
Ureteric fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (6) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 13 (15) | 15 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 9 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5) | 7 (9) | 6 (7)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 15 (17) | 17 (17) | 17 (17)
Hypotension (Vascular disorders) | 0 (0) | 4 (4) | 4 (4)
Lymphedema (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 7 (9) | 7 (7) | 4 (4)
Vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Paclitaxel) (N=272) | Arm B (Nab-paclitaxel) (N=264) | Arm C (Ixabepilone) (N=238)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood disorder (Blood and lymphatic system disorders) | 1 (4) | 2 (5) | 2 (4)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 3 (6) | 1 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 49 (202) | 49 (165) | 40 (128)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (3) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 3 (5) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 2 (4) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (20) | 3 (7) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (2) | 3 (5)
Cushingoid (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (28) | 2 (3) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 2 (4) | 3 (3)
Eye disorder (Eye disorders) | 2 (2) | 4 (5) | 0 (0)
Flashing vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 4 (12) | 13 (31) | 2 (3)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 2 (2) | 9 (19) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (4) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (13) | 7 (10) | 10 (12)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (4) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 35 (84) | 36 (95) | 45 (87)
Diarrhea (Gastrointestinal disorders) | 35 (74) | 36 (67) | 45 (85)
Dry mouth (Gastrointestinal disorders) | 3 (6) | 3 (4) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 11 (20) | 13 (19) | 20 (34)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 3 (4) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (3) | 5 (6) | 5 (6)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 5 (11) | 1 (1) | 3 (5)
Gastroscopy abnormal (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 2 (5) | 1 (1) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 (5) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 3 (3) | 2 (6) | 8 (15)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 21 (35) | 22 (40) | 16 (32)
Nausea (Gastrointestinal disorders) | 48 (92) | 52 (123) | 75 (160)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (9)
Oral pain (Gastrointestinal disorders) | 2 (2) | 4 (10) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (11)
Peritoneal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 9 (24) | 8 (11) | 5 (8)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Tooth development disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 18 (24) | 27 (45) | 29 (48)
Chest pain (General disorders) | 6 (11) | 2 (2) | 3 (3)
Chills (General disorders) | 2 (2) | 4 (7) | 4 (5)
Edema limbs (General disorders) | 11 (37) | 13 (37) | 11 (46)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 208 (1397) | 213 (1186) | 205 (1036)
Fever (General disorders) | 4 (5) | 5 (6) | 7 (14)
Flu-like symptoms (General disorders) | 1 (1) | 2 (2) | 1 (1)
Gait abnormal (General disorders) | 0 (0) | 1 (2) | 0 (0)
General symptom (General disorders) | 1 (4) | 2 (4) | 2 (3)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 3 (5)
Localized edema (General disorders) | 4 (13) | 1 (2) | 2 (2)
Pain (General disorders) | 21 (34) | 13 (16) | 12 (24)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (5) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 23 (32) | 28 (48) | 17 (19)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 3 (7) | 3 (5) | 2 (2)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1) | 2 (2)
Catheter related infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (7) | 0 (0) | 2 (3)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 8 (9) | 6 (7) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Nail infection (Infections and infestations) | 2 (2) | 3 (5) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 6 (7) | 6 (7) | 3 (6)
Skin infection (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 5 (5) | 4 (5) | 6 (6)
Ureteritis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (12) | 6 (6) | 9 (14)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Intraoperative breast injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 10 (28) | 10 (32) | 9 (15)
Alanine aminotransferase increased (Investigations) | 14 (18) | 18 (28) | 18 (35)
Alkaline phosphatase (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 11 (31) | 11 (27) | 18 (31)
Aspartate aminotransferase increased (Investigations) | 15 (21) | 18 (31) | 17 (39)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 4 (6)
Creatinine increased (Investigations) | 9 (16) | 4 (7) | 2 (14)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
INR increased (Investigations) | 2 (3) | 3 (6) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 1 (1) | 6 (9)
Leukocyte count decreased (Investigations) | 55 (188) | 87 (242) | 41 (98)
Lymphocyte count decreased (Investigations) | 7 (26) | 10 (27) | 5 (13)
Neutrophil count decreased (Investigations) | 116 (447) | 178 (650) | 64 (144)
Platelet count decreased (Investigations) | 23 (50) | 28 (65) | 16 (44)
Serum cholesterol increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Weight gain (Investigations) | 3 (9) | 0 (0) | 3 (6)
Weight loss (Investigations) | 11 (19) | 13 (35) | 14 (31)
Anorexia (Metabolism and nutrition disorders) | 24 (50) | 25 (48) | 30 (61)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (2) | 3 (7) | 1 (6)
Blood glucose increased (Metabolism and nutrition disorders) | 32 (129) | 29 (64) | 29 (64)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 7 (9) | 6 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 10 (17) | 8 (19) | 11 (23)
Serum calcium decreased (Metabolism and nutrition disorders) | 9 (18) | 8 (12) | 10 (16)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 11 (21) | 9 (15) | 12 (21)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (15) | 3 (3) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 11 (33) | 10 (19) | 14 (25)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 (122) | 38 (75) | 37 (117)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (28) | 12 (33) | 26 (51)
Bone pain (Musculoskeletal and connective tissue disorders) | 20 (41) | 11 (21) | 13 (30)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (5) | 2 (2)
Fibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (9) | 9 (19) | 3 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 2 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (9) | 1 (2) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 92 (336) | 99 (295) | 77 (210)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (3) | 3 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (7) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (27) | 9 (12) | 11 (21)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 3 (4) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 13 (20) | 11 (14) | 15 (27)
Dysgeusia (Nervous system disorders) | 12 (61) | 15 (40) | 29 (59)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 20 (28) | 22 (43) | 30 (50)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (4) | 3 (3) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (5)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 46 (110) | 66 (208) | 47 (204)
Peripheral sensory neuropathy (Nervous system disorders) | 216 (1533) | 206 (1320) | 175 (1043)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 5 (5) | 1 (1) | 4 (4)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Agitation (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 16 (29) | 7 (11) | 10 (19)
Confusion (Psychiatric disorders) | 2 (4) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 13 (33) | 14 (20) | 14 (33)
Euphoria (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 18 (41) | 13 (25) | 19 (35)
Libido decreased (Psychiatric disorders) | 1 (4) | 1 (1) | 1 (8)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder hemorrhage (Renal and urinary disorders) | 2 (5) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (2)
Cystitis (Renal and urinary disorders) | 3 (4) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin urine positive (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 3 (5) | 3 (4) | 2 (3)
Kidney pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 58 (211) | 64 (188) | 50 (125)
Ureteric hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urethral hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (7) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 5 (6) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 2 (2) | 3 (5) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 2 (4) | 2 (3)
Irregular menstruation (Reproductive system and breast disorders) | 2 (7) | 0 (0) | 0 (0)
Ovulation pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 3 (4) | 1 (1) | 2 (6)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (5)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2) | 5 (5) | 2 (5)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 7 (10) | 14 (22)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (65) | 20 (43) | 24 (54)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27 (62) | 29 (61) | 36 (91)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 68 (174) | 56 (185) | 47 (112)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (9) | 2 (2)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 9 (19) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 5 (9) | 5 (12)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7) | 4 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 7 (9) | 6 (8)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 3 (7) | 6 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 35 (151) | 26 (65) | 40 (116)
Chest wall necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (7) | 7 (10)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 5 (16) | 7 (15) | 2 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 32 (96) | 24 (63) | 16 (28)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 8 (19) | 4 (17)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (11) | 3 (6)
Rash desquamating (Skin and subcutaneous tissue disorders) | 17 (28) | 34 (71) | 14 (33)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 11 (17) | 5 (6) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (15) | 4 (10) | 1 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (6) | 2 (4) | 2 (4)
Sweating (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (8) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 3 (4) | 3 (3) | 2 (2)
Hot flashes (Vascular disorders) | 5 (15) | 9 (12) | 10 (25)
Hypertension (Vascular disorders) | 127 (596) | 97 (418) | 90 (345)
Hypotension (Vascular disorders) | 1 (1) | 4 (4) | 5 (6)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (18) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 7 (30) | 8 (13) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less